CLINICAL TRIAL: NCT06137976
Title: Surgeon Perception of Gastric Decompression at Time of Gynecologic Laparoscopy, a Randomized Control Trial
Brief Title: Surgeon Perception of Gastric Decompression at Time of Gynecologic Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Chief of Minimally Invasive Gynecologic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU00219580
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Surgical Procedures; Gastric Injury; Aspiration; Nausea, Postoperative; Postoperative Complications; Enhanced Recovery After Surgery; Laparoscopy
Keywords: Gastric decompression; Gynecologic surgery; Gynecologic laparoscopy; Surgical visualization; Enhanced Recovery After Surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: * Block randomization in groups of 10 to either receive nasogastric or orogastric intubation after endotracheal intubation prior to abdominal entry for the duration of the surgery or no gastric decompression at all.
  * Sequentially numbered, opaque, sealed envelope (SNOSE) technique
Who Masked: Participant, Care Provider
Masking Description: * Patient will masked to group assignment and will be under anesthesia during intervention.
  * Surgeon will be masked to group assignment. Placement of the nasogastric or orogastric tube will occur while the surgeon is scrubbing and out of the room. There will be a drape over the face until the surgical drapes are covering the patient to maintain surgeon blinding. Removal of tube will take place prior to undraping the patient to maintain blinding.
  * All documents noted group assignment will be in an opaque envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric decompression (Experimental): Placement of the nasogastric or orogastric tube will occur after intubation while surgeons are scrubbing and out of the room to maintain blinding. At the end of surgery, the nasogastric or orogastric tube will be removed prior to removal of the surgical drapes to ensure the surgeon remains blinded. Patients will then be returned to routine post-operative care as otherwise planned or necessitated by surgery.
  Interventions: Procedure: Gastric decompression (oropharyngeal or nasopharyngeal gastric tube)
- No gastric decompression (No Intervention): No placement of gastric decompression tube.

INTERVENTIONS:
Procedure: Gastric decompression (oropharyngeal or nasopharyngeal gastric tube) — Placement of tube through the nose or mouth into the stomach for gastric decompression
  Arms: Gastric decompression

SUMMARY:
The goal of this clinical trial is to test whether it is necessary to decompress the stomach during gynecologic laparoscopy.

The main questions it aims to answer are:

* Is there appropriate visualization during surgery without stomach decompression?
* Can the surgeon tell the stomach is decompressed?
* Is the stomach at risk for injury during surgery?
* How is the patient's postoperative experience affected?

Participants will undergo their planned surgery as usual and will be asked to complete log about their recovery for the first week after surgery.

Researchers will compare patients who have their stomach decompressed during surgery to those who do not undergo stomach decompression to see if it is necessary.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) pathways are a framework for management before, during, and after surgery that has demonstrated several benefits from a cost, complication, and satisfaction standpoint. In the field of gynecologic surgery, the American College of Obstetricians and Gynecologists (ACOG) recommends utilization of these pathways with particular emphasis on the importance of implementation of multiple components together. A literature review of 47 ERAS programs specific to obstetrics and gynecology (requiring at least four individual components of ERAS for inclusion) overall supported its use, however, recommended randomized control trials to evaluate each component of the pathway.

One component of the ERAS pathway includes gastric decompression in the perioperative setting. In 1999, before the advent of ERAS, an anesthesiologist recommended routine use of intraoperative gastric decompression to reduce risk of gastric perforation, citing laparoscopic general surgery anesthesia recommendations from 1993. The general surgery paper highlights the possibility for unintentional gastric distention with mask ventilation prior to anesthesia induction with associated increased risk of trocar injury, however, does not discuss incidence or rates of this phenomena. There is discussion of an association with increased intraabdominal pressure and regurgitation of gastric contents, however, nasogastric decompression is not addressed within this context.

Indications for nasogastric tube use in general include treatment of ileus, administration of medications, enteral nutrition, and stomach lavage. Currently available anesthesia recommendations include routine use of gastric tubes during induction with general endotracheal anesthesia. Importantly, it is noted that gastric drainage or suction does not remove particulate matter or guarantee full emptying. In fact, one study looking at use of nasogastric intubation after induction of anesthesia found that patients who underwent nasogastric intubation had significant gastroesophageal reflux disease in the perioperative period and a reduced ability to clear refluxed acid from the distal esophagus. Several other studies examining the routine placement of a nasogastric tube following abdominal surgery also found that patients who underwent gastric decompression had higher rates of fever, pneumonia, and other pulmonary complications. In these studies, those with a nasogastric tube had lower rates of emesis, but increased patient discomfort, no significant difference in the rates of nausea, and longer time to return of bowel function. One comparative study from the general surgery literature evaluating nasogastric decompression during open abdominal surgeries included a subgroup without placement at all in the perioperative period. This subgroup demonstrated significantly less events of atelectasis, fever, and patient discomfort. Furthermore, the routine use of gastric decompression is not benign, and some evidence suggests the benefits of routinely avoiding nasogastric intubations outweigh the risks.

Data has shown that early post-operative nasogastric tube discontinuation (including prior to transfer to post-anesthesia care) is associated with faster return to bowel function and decreased rates of postoperative ileus, as well as decreased hospital stay and rates of pulmonary complications. While it is commonplace for recommended ERAS diet status leading up to and after surgery in most institutions, (i.e., elimination of mechanical bowel prep, removal of nasogastric decompression prior to extubation), there is no clinical evidence available to date on utilization of intraoperative gastric decompression specifically for gynecologic laparoscopic cases.

Additionally, nasogastric or orogastric tubes may contribute to high costs of the operating room. On average, a nasogastric tube costs on average 4 dollars and seventy-five cents (based on cost for pack of 10) at this institution according to 2023 supply invoices. In 2022, a call to action in the Journal of Minimally Invasive Gynecologic Surgery urged gynecologic surgeons to consider their role in safe and green practices in the operating room. Evaluating use of routine gastric decompression at time of gynecologic surgery is an opportunity to decrease potential costs and environmental impact.

Within the field of gynecologic oncology, recommendations are against routine nasogastric intubation and for early post-operative removal prior to extubation, however, possible reduction of risk of injury associated with Veress needle or trocar entry are noted. Regarding minimally invasive gynecologic surgery recommendations specifically, the first guidelines in 2020 discussed that patients with normal gastric emptying may intake up to 400 milliliters of clear liquids up to 2 hours prior to anesthesia with an equivalent gastric volume to overnight fasting. Nasogastric decompression was not recommended for prevention of post-operative nausea and vomiting; however, its use was not discussed in terms of prevention of entry injury or prevention of postoperative pneumonia.

Overall, gastric injury is a rare complication of gynecologic surgery estimated to occur less than 0.5% of the time. A systematic review of 28 articles assessed the location and mechanism of gastric injury at the time of gynecologic surgery by analyzing 42 injuries. In the study, 93% of gastric injuries occurred upon entry with the Veress needle, which was used in 79% of cases. There was only one case with nasogastric decompression prior to entry and the location of entry was the left upper quadrant as opposed to the umbilicus.

Given rarity of gastric injury at time of laparoscopic gynecologic surgery and limited to no data regarding purported benefit of intraoperative gastric decompression, particularly regarding reduction of trocar injury rates, its routine use should be examined. Routine use may be associated with harmful potential for post-operative complications including pneumonia, delayed bowel function, and patient discomfort. In 2014, a similar evaluation of routine mechanical bowel preparation at time of laparoscopic hysterectomy demonstrated no difference in surgeon perception of visualization and ability to complete the procedure safely with or without mechanical bowel preparation. Similarly, the paper recognizes the purported benefits of routine mechanical bowel preparation to be largely untested prior to this study and the potential association for harm with patient discomfort and risks without improved surgical outcomes with existing data derived from laparotomies. When examined, both the primary and assistant surgeon had moderate agreement and accurately assessed preoperative bowel preparation a little more than half of the time, indicating that surgeon perception may not be reflective of perioperative measures.

The aim of this study is to examine the routine use of intraoperative gastric decompression during gynecologic laparoscopy. The primary outcome is surgeon perception of visualization of gastric decompression and surgery characteristics. Secondary outcomes are factors associated with patients' post-operative experience such as nausea and vomiting, return of bowel function, and naso- and oro-pharyngeal discomfort. The investigators hypothesize that limiting gastric decompression for specific medical indications as opposed to routine use will not be associated with an increased risk of harm such as gastric injury and poor surgical visualization for gynecologic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gynecologic laparoscopy for the following indications: hysterectomy, adnexal surgery, benign and malignant tumors or disease, diagnostic purposes, lysis of adhesions, and pelvic pain.
* Surgery being performed by gynecologic surgeon with or without minimally invasive gynecologist certification, gynecologic oncologists, urogynecologists, and reproductive endocrinologists.

Exclusion Criteria:

* Entry sites other than umbilical
* Planned or high suspicion for bowel surgery
* Anticipated surgical time >4 hours
* Known diagnosis of gastric reflux disease or peptic ulcer disease
* Prior history of gastric or esophageal surgery excluding endoscopy
* Day of surgery emesis events
* Difficult intubation determined by anesthesia
* Intrauterine pregnancy
* Chronic lung disease
* Individuals with smoking history.
* Individuals who do not speak English due to limitations in ability to reliably obtain informed consent in their primary language.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Adequate gastric decompression | At time of surgery
  The primary endpoint is the percentage of cases rated as adequate decompression by the surgeon.
Gastric injury | Up to six weeks post-operatively
  The primary safety endpoint is the estimated negligible rate of gastric injury.

SECONDARY OUTCOMES:
Presence of gastric decompression tube | At time of surgery
  Accurate determination of presence of orogastric or nasogastric tube via intraoperative survey
Gastric injury risk assessment | At time of surgery
  Percentage of cases in which the surgeon believes the stomach was at risk for injury during umbilical entry
Degree of stomach decompression | At time of surgery
  Perceived degree of stomach decompression, rated qualitatively as "excellent," "good," "fair," or "poor"
Entry proximity | At time of surgery
  Estimated distance between the umbilicus and stomach on abdominal entry
Post-operative experience questionnaire | First 7 days after surgery
  Patients' postoperative experience including rates of nausea and vomiting, nasal, and oropharyngeal discomfort, and time to return of bowel function as measured by a patient reported symptom log
Post-operative complications | Up to six weeks post-operatively
  A secondary safety endpoint is rates of postoperative complications which may be related to gastric decompression including aspiration or pneumonia as measured by electronic medical record chart review post operatively.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - 259 E Erie - Northwestern, Chicago, Illinois
  - Prentice Women'S Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkow, L. Rapid sequence induction and intubation (RSII) for anesthesia. UpToDate, 2023. https://www.uptodate.com/contents/rapid-sequence-induction-and-intubation-rsii-for-anesthesia
- [Background] Cheatham ML, Chapman WC, Key SP, Sawyers JL. A meta-analysis of selective versus routine nasogastric decompression after elective laparotomy. Ann Surg. 1995 May;221(5):469-76; discussion 476-8. doi: 10.1097/00000658-199505000-00004. PMID 7748028
- [Background] Chui PT, Gin T, Oh TE. Anaesthesia for laparoscopic general surgery. Anaesth Intensive Care. 1993 Apr;21(2):163-71. doi: 10.1177/0310057X9302100205. PMID 8517506
- [Background] Coskun F. Anesthesia for gynecologic laparoscopy. J Am Assoc Gynecol Laparosc. 1999 Aug;6(3):245-58. doi: 10.1016/s1074-3804(99)80057-7. PMID 10459023
- [Background] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Background] Hodin, R. Inpatient placement and management of nasogastric and nasoenteric tubes in adults. UpToDate, 2023. https://www.uptodate.com/contents/inpatient-placement-and-management-of-nasogastric-and-nasoenteric-tubes-in-adults
- [Background] Hu H, Choi JDW, Edye MB, Aitken T, Kapurubandara S. Gastric Injury at Laparoscopy for Gynecologic Indications: A Systematic Review. J Minim Invasive Gynecol. 2022 Nov;29(11):1224-1230. doi: 10.1016/j.jmig.2022.09.058. Epub 2022 Sep 30. PMID 36184063
- [Background] Manning BJ, Winter DC, McGreal G, Kirwan WO, Redmond HP. Nasogastric intubation causes gastroesophageal reflux in patients undergoing elective laparotomy. Surgery. 2001 Nov;130(5):788-91. doi: 10.1067/msy.2001.116029. PMID 11685187
- [Background] Michowitz M, Chen J, Waizbard E, Bawnik JB. Abdominal operations without nasogastric tube decompression of the gastrointestinal tract. Am Surg. 1988 Nov;54(11):672-5. PMID 3190004
- [Background] Nelson R, Edwards S, Tse B. Prophylactic nasogastric decompression after abdominal surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD004929. doi: 10.1002/14651858.CD004929.pub3. PMID 17636780
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Rao W, Zhang X, Zhang J, Yan R, Hu Z, Wang Q. The role of nasogastric tube in decompression after elective colon and rectum surgery: a meta-analysis. Int J Colorectal Dis. 2011 Apr;26(4):423-9. doi: 10.1007/s00384-010-1093-4. Epub 2010 Nov 24. PMID 21107848
- [Background] Scheib SA, Thomassee M, Kenner JL. Enhanced Recovery after Surgery in Gynecology: A Review of the Literature. J Minim Invasive Gynecol. 2019 Feb;26(2):327-343. doi: 10.1016/j.jmig.2018.12.010. Epub 2018 Dec 20. PMID 30580100
- [Background] Schwartz KM, Wright KN, Richards EG, King LP, Park AJ. Sustainability in Healthcare: A Call to Action for Surgeons and Healthcare Leaders. J Minim Invasive Gynecol. 2022 Sep;29(9):1040-1042. doi: 10.1016/j.jmig.2022.06.024. Epub 2022 Jul 1. No abstract available. PMID 35788396
- [Background] Siedhoff MT, Clark LH, Hobbs KA, Findley AD, Moulder JK, Garrett JM. Mechanical bowel preparation before laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2014 Mar;123(3):562-567. doi: 10.1097/AOG.0000000000000121. PMID 24499763
- [Background] Stone R, Carey E, Fader AN, Fitzgerald J, Hammons L, Nensi A, Park AJ, Ricci S, Rosenfield R, Scheib S, Weston E. Enhanced Recovery and Surgical Optimization Protocol for Minimally Invasive Gynecologic Surgery: An AAGL White Paper. J Minim Invasive Gynecol. 2021 Feb;28(2):179-203. doi: 10.1016/j.jmig.2020.08.006. Epub 2020 Aug 20. PMID 32827721
- [Result] ACOG Committee Opinion No. 750 Summary: Perioperative Pathways: Enhanced Recovery After Surgery. Obstet Gynecol. 2018 Sep;132(3):801-802. doi: 10.1097/AOG.0000000000002819. PMID 30134419

DOCUMENTS (1):
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT06137976/ICF_000.pdf